CLINICAL TRIAL: NCT00247338
Title: Comparing With Traditional Nitrogen Calorie Parenteral Nutrition Support, the Impact of Low Calorie and Low Nitrogen Intake on the Clinical Outcome of Gastrointestinal Postoperative Patients, Multicentre Post-Marketing Clinical Study
Brief Title: The Impact of Low Calorie and Low Nitrogen Parenteral Nutrition Support on the Clinical Outcome of Postoperative Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sino-Swed Pharmaceutical Corporation (Industry)
Collaborators: Guangzhou S Y S Medical School hospital (Unknown); Wuhan TongJi Hospital (Other); Beijing 301 hospital (Unknown); Jie-Ping Wu Medical Foundation (Unknown)
Responsible Party: ZM Jiang, Peking Union Medical Hospital
Organization: Fresenius Kabi Sino-Swed Pharmaceutical Corp. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypocaloric PN
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Gastrointestinal Neoplasms; Postoperative Complications
Keywords: parenteral nutrition; low calorie; low nitrogen; gastrointestinal neoplasms; gastrointestinal diseases; gastrectomy; colectomy; rectectomy; operations
MeSH Terms: conditions — Gastrointestinal Neoplasms; Postoperative Complications; Hyperphagia; Gastrointestinal Diseases

INTERVENTIONS:
Drug: low calorie, low nitrogen parenteral nutrition for patient with NRS score 3

SUMMARY:
The study is designed to investigate the influence of parenteral nutrition (PN) with low nitrogen and calorie supply on the clinical outcome of patients after an operation compared to that of traditional PNs.

DETAILED DESCRIPTION:
Wretlind from Sweden invented fat emulsion as early as 1961, which has been applied to parenteral nutrition. Dudrick and Wilmore from America introduced intravenous nutrition containing carbohydrates and amino acids, which was termed as high intravenous nutrition in 1967. Afterwards, it was proven that this treatment cannot improve clinical outcome but increases complications, such as infection, etc. Because of the action of catecholamine and corticosteroids under stress after an operation, insulin resistance becomes a main indicator of endocrine problems for patients. Under such circumstances, even intake of glucose at physiological doses can result in hyperglycosemia and increase the incidence of complications of infection and metabolism. Overseas and domestic scholars studied parenteral nutrition (PN) with low nitrogen and calorie supply long ago, and the results revealed that PN with low nitrogen and calorie supply can significantly decrease oxygen consumption of patients under stress of an operation, alleviate the inflammation response, reduce the rate of cholestasis and cut the treatment cost during hospitalization. On the other hand, catabolism of protein significantly increases after operation and trauma, but it cannot be simply corrected by high dose amino acid intake. Contrarily, improperly increasing of the intake of amino acids aggravates metabolism further. A domestic study on PN with a low calorie supply has revealed benefits on the clinical outcome of patients after an operation, such as a domestic randomised controlled study that has proven that intravenous nutrition with a low nitrogen and calorie supply significantly lowered the level of blood glucose, cut nutrition related medicine costs, shortened the length of hospital stay and reduced the incidence of phlebitis after operation, and also has the tendency to reduce the incidence of complications after an operation. Meta analysis has revealed that PN with a low nitrogen and calorie supply can control blood glucose better and may reduce the incidence of infection related complications, and has the tendency of shortening the length of hospital stay.

The development of all-in-one PN has experienced the process of sequential single bottle infusion, poly-bottle serial infusion, hospital prepared all-in-one solution and industrialized three compartment bags, and currently, the utilization of industrialized three compartment bags has been the dominant tendency of clinical parenteral nutrition among countries in Europe and Asia. Domestically Kabiven peripheral (FK, Germany, 1440 ml H20040008, 1920 ml H20040019) are the first three compartment bags, which is a pre-filling standard all-in-one nutrition solution. The two specifications (1440 ml,1920 ml) first launched to the market already satisfy most demands of PN support for patients, and provide PN with a low nitrogen and calorie supplying administration platform for patients after operation, spare time for the preparation of all-in-one nutrition solution, and avoid preparing such solutions under the common clean condition in hospitals.

Up to now, there is no report of a randomized controlled study about the utilization of three compartment bags domestically.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone resection of stomach, intestine, or rectum, having the indication of nutrition
* Nutrition risk screening scores around 3
* The age of the patients must be between 18 to 80
* The patients sign the confirmed consent letter
* Weight falls in the range of either 45-56 kg or 60-75 kg

Exclusion Criteria:

* Pregnant or breast feeding
* Contraindication of fluid infusion, acute pulmonary edema, brain edema and functional insufficiency of the heart
* Hypersensitive to the ingredient of the trial product nutrient
* Chemotherapy within 7 days before the beginning of this trial
* Unstable angina pectoris
* Diabetes mellitus
* Disorder of lipid metabolism: triglycerides, cholesterol increased by 1.5 times above the reference value
* Abnormal renal function: serum creatinine or BUN 1.5 times above normal reference value
* Abnormal liver function: ALT or serum total bilirubin 1.5 times above normal reference value
* Having severe drug allergy history and/or asthma
* On operation day, blood loss above 800 ml
* Contraindication to parenteral nutrition
* Receiving regular parenteral nutrition within 7 days before the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-04; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Infectious complications | POD+1 to POD+14

SECONDARY OUTCOMES:
Systemic inflammatory response syndrome | POD+1 to POD + 7
The length of hospital stay after operation | POD+1 to discharge
Post-operative nutritional cost & total treatment cost | POD+1 to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Wen-hua Zhan, MD,FACS, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Zhu-Ming Jiang, MD, FACS, Study Chair — Parenteral & Enteral Centre, Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Department of Gastrointestinal Surgery, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Department of General Surgery, Affiliated Hospital of Medical University of Tongji, Wuhan, Hubei
  - Department of General Surgery, General Hospital of PLA, Beijing

REFERENCES:
- [Derived] Zhan WH, Jiang ZM, Tang Y, Wu YP, Liu JW, Zhang YJ, Chen W, Liu T, Yao C. [Impact of hypocaloric and hypo-nitrogen parenteral nutrition on clinical outcome in postoperative patients: a multi-center randomized controlled trial of 120 cases]. Zhonghua Yi Xue Za Zhi. 2007 Jul 3;87(25):1729-33. Chinese. PMID 17919374